CLINICAL TRIAL: NCT05637320
Title: Biobehavioural Regulation of Negative Emotion as a Transdiagnostic Mechanism of Children's Psychotherapy
Brief Title: Big Feelings: A Study on Children's Emotions in Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Centre for Addiction and Mental Health (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Kristel Thomassin, Associate Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 004-2022
Record Dates: First submitted 2022-11-15; First posted 2022-12-05 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Anxiety Disorders; Depressive Disorder; Mood Disorders; Conduct Disorder; Oppositional Defiant Disorder; Regulation, Emotion; Child Behavior Disorders; Trauma and Stressor Related Disorders
Keywords: Child psychotherapy; Emotion regulation; Physiology; Mechanism of change
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Mood Disorders; Conduct Disorder; Oppositional Defiant Disorder; Emotional Regulation; Child Behavior Disorders; Trauma and Stressor Related Disorders

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial, consisting of an intervention arm and a control arm, which will occur concurrently. Participants will be continually enrolled in the study until 202 parent-child dyads are recruited.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Treatment will be administered to participants in this arm.
  Interventions: Behavioral: Modular Approach to Therapy for Children with Anxiety, Depression, Trauma or Conduct Problems
- Control Arm (No Intervention): No treatment will be administered to participants in this arm until post-test assessment has been completed.

INTERVENTIONS:
Behavioral: Modular Approach to Therapy for Children with Anxiety, Depression, Trauma or Conduct Problems — The intervention arm will consist of a transdiagnostic psychotherapy program: The Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, or Conduct Problems (MATCH-ADTC). MATCH draws from various domains of evidence-based treatment and consists of 33 treatment modules. There are several core module sequences for problem areas such as depression, anxiety, trauma, and disruptive behavior, and a clinician can utilize these sequences based on the primary concern of the presenting child. If an individual reports additional stressors or comorbid conditions, the clinician can modify the sequence of the modules to address these comorbidities. MATCH treatment is flexible and is tailored for each individual client.
  Other Names: MATCH-ADTC
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to learn about how psychotherapy works for children and adolescents aged 8 - 15 with anxiety, depression, trauma, or disruptive behaviour. The main question it aims to answer is:

• Is the biobehavioural regulation of negative emotion a transdiagnostic mechanism of treatment response in psychotherapy for children with anxiety, depression, trauma and/or disruptive behaviour?

Children and their parents will be randomly assigned to an evidence-based, transdiagnostic treatment (the Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, and Conduct Problems; MATCH-ADTC) or a waitlist control condition. Participants in both groups will complete a baseline assessment, weekly measures consisting of brief symptom scales and medication tracking, and quarterly assessments every 3 months. Following the intervention/waitlist period, our team will conduct post-test assessments. All assessments, except for the weekly surveys, will consist of symptom scales, clinical interviews, experimental tasks and physiological measures.

DETAILED DESCRIPTION:
Research shows that evidence-based psychotherapies for children's mental health problems are only moderately effective, and as many as 50% of children will fail to respond to treatment or will drop out of treatment. There is thus significant room for improvement. One way to improve outcomes for children and their families is to understand how psychotherapy works for children and to make personalized adjustments to optimize their effectiveness.

The primary aim of this study is to test biobehavioural regulation of negative emotion as a transdiagnostic mechanism of treatment response in psychotherapy for children with anxiety, depression, trauma, and/or disruptive behavior. Treatment response will be evaluated as pre-to-post change in symptoms and the rate of symptom change. Biobehavioural regulation of emotion will be measured using a multimodal approach comprising validated parent and child-report questionnaires, performance on behavioral and cognitive regulation tasks, and physiological reactivity. Our second aim is to apply association rule mining, a machine learning technique, to uncover patterns governing variations in regulation components throughout the course of treatment. Patterns will be expressed in the form of data-driven and rule-based algorithms reflecting the relation between emotion regulation and treatment response.

Clinicians will be trained on administering the Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, and Conduct Problems (MATCH-ADTC) treatment.

Children aged 8 - 15 seeking psychotherapy for anxiety, depression, trauma, or disruptive behaviour will be recruited from two outpatient mental health clinics. Approximately 202 dyads of a child and parent will be recruited for this study. Participants will be randomly assigned to the intervention arm or the waitlist control arm. Participants in both groups will complete a baseline assessment, weekly measures consisting of brief symptom scales and medication tracking, and quarterly assessments every 3 months. Following the intervention/waitlist period, our team will conduct post-test assessments. All assessments, except for the weekly surveys, will consist of symptom scales, clinical interviews, experimental tasks and physiological measures.

ELIGIBILITY:
Inclusion Criteria:

* Child must be between the ages of 8 and 15 years old and have English proficiency
* Parents must be over the age of 18 and have English proficiency
* Must be seeking psychosocial treatment for concerns related to anxiety, depression, or disruptive behaviours

Exclusion Criteria:

* Child has low cognitive functioning that would prevent active participation in research tasks
* Child reports active suicidality that requiring acute care or hospital intervention
* Child meets criteria for psychosis, schizophrenia spectrum disorders, eating disorders or autism spectrum disorders
* Child does not assent to participate in the study

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 202 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in parent-rated child psychopathology symptoms | Change at quarterly (3 month intervals after pre-test), change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured through the Child Behavior Checklist (CBCL), a 113-item measure of child psychopathology symptoms that is completed by parents (parent-report). Parents will rate items on a three-point Likert scale from (0 = Never, 1 = Sometimes, 2 = Often) with scores across syndrome scales (anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behaviour, and aggressive behaviours) and DSM-oriented scales (affective problems, anxiety problems, somatic problems, attention-deficit/hyperactivity problems, oppositional defiant problems, and conduct problems).
Change in child self-reported psychopathology symptoms | Change at quarterly (3 month intervals after pre-test), change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured through the Youth Self Report (YSR) a 112-item measure of child psychopathology symptoms that is completed by children aged 11 - 15 (youth-report). Children will rate items on a three-point Likert scale from (0 = Never, 1 = Sometimes, 2 = Often) with scores across syndrome scales (anxious/depressed, withdrawn/depressed, somatic problems, social problems, thought problems, rule-breaking behaviour, and aggressive behaviours) and DSM-oriented scales (depressive problems, anxiety problems, somatic problems, attention-deficit/hyperactivity problems, oppositional defiant problems, and conduct problems).
Change in child psychopathology symptoms (past week) | Change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured through the Behavior and Feelings Survey (BFS), a 12-item measure of child psychopathology symptoms to be completed by parents (parent-report) and children (youth-report). Parents and children will rate items on a five-point Likert scale from 0 (Not a problem) to 4 (A very big problem) with greater scores (internalizing subscale range = 0-24; externalizing subscale range = 0-24; total score range = 0-48) indicating more severe psychopathology. The BFS generates Internalizing, Externalizing, and Total Problems scores.
Change in child emotional-behavioural problems | Change at quarterly (3 month intervals after pre-test), change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured through the Top Problems Assessment (TPA), a brief, clinical interview that is completed by parents (parent-report) and children (youth-report). Children and parents will identify and describe one to three primary issues, rate the severity of each problem on a scale of 0 (not a problem) to 4 (a very big problem). They will then rank order the problems from 1 (biggest problem) to 3 (least big problem).
Change in child impairment | Change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured through the Brief Impairment Scale (BIS), a 23-item measure of child impairment that is completed by one or both parents (parent-report). Parents will rate items on a four-point Likert scale from 0 (No problem) to 3 (A Serious Problem) with greater scores across three domains (interpersonal subscale = 0 - 24, school/work = 0 - 24, self-fulfillment = 0 - 24) indicating more severe impairment.
Change in ratings of child emotion regulation | Change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured through the Negative Emotionality subscale of the Child and Adolescent Dispositions Scale (CADS), a scale of child emotion regulation to be completed by parents (parent-report) and children (youth-report for children). Parents and children will rate the items on a four-point Likert scale from 1 (Not at all) to 4 (Very much/very often) with greater scores (range = 7 - 28) indicating poorer emotion regulation.
Change in child physiological emotion regulation (heart rate variability) | Change at quarterly (3 month intervals after pre-test), change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured by child heart rate variability during the completion of lab tasks (Modified Trier Social Stress Test for Children, Piñata Task, Cognitive Reappraisal, Parent-Child Conflict Discussion).
Change in child physiological emotion regulation (skin conductance) | Change at quarterly (3 month intervals after pre-test), change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome measure will be measured by child skin conductance level during the completion of lab tasks (Modified Trier Social Stress Test for Children, Piñata Task, Cognitive Reappraisal, Parent-Child Conflict Discussion).

SECONDARY OUTCOMES:
Change in child psychopathology symptoms on a weekly basis | From pre-test assessment to post-test assessment, an average of 4 - 6 months
  This outcome will be measured through the Behavior and Feelings Survey (BFS), a 12-item measure of child psychopathology symptoms to be completed by parents (parent-report) and children (youth-report). Parents and children will rate items on a five-point Likert scale from 0 (Not a problem) to 4 (A very big problem) with greater scores (internalizing subscale range = 0-24; externalizing subscale range = 0-24; total score range = 0-48) indicating more severe psychopathology
Change in child emotion regulation on a weekly basis | From pre-test assessment to post-test assessment, an average of 4 - 6 months
  This outcome will be measured through the Negative Emotionality subscale of the Child and Adolescent Dispositions Scale (CADS), a scale of child emotion regulation to be completed by parents (parent-report) and children (youth-report). Parents and children will rate the items on a four-point Likert scale from 1 (Not at all) to 4 (Very much/very often) with greater scores (range = 7 - 28) indicating poorer emotion regulation.
Change in parent psychopathology symptoms | Change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured through the Brief Symptom Inventory (BSI-18), an 18-item measure of adult psychopathology symptoms to be completed by parents (parent-report). Parents will rate items on a five-item Likert scale from 0 (Not at all) to 4 (Extremely) with greater scores on three dimensions (somatization, depression, anxiety, total score range = 0 - 72) indicating more severe psychopathology.
Change in parent stress | Change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured through the Parenting Stress Index-Short form (PSI-SF), a 36-item of stress in the parent-child relationship. Parents will rate items on a five-point Likert scale from 1 (Strongly Disagree) to 5 (Strongly Agree) with scores categorized into subscales (parental distress, parent-child dysfunctional interaction, and difficult child), and higher scores (range = 0 - 180) indicating greater stress.
Change in parent emotion regulation | Change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured through the Difficulties in Emotion Regulation Scale - Short Form (DERS), an 18-item self-report measure of emotion regulation difficulties to be completed by parents. Parents will indicate the frequency with which they experience difficulties with emotion regulation on a five-point Likert scale from 1 (Almost never) to 5 (Almost always), with greater total scores (range = 18 - 90) indicating greater difficulties with emotion regulation.
Change in family function | Change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured through the Family Functioning Style Scale (FFSS), a 26-item self-report measure of family function to be completed by parents. Parents will rate items on a five-point Likert scale from 0 (Not at all like my family) to 4 (Almost always like my family), with scores categorized into five subscales (interactional patterns, family values, coping strategies, family commitment and resource mobilization) of a family's functioning style
Change in family organization | Change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured using the Confusion, Hubbub, and Order Scale (CHAOS), a 15-item measure of family organization within the home, with 7 items reflecting routine and organization and 8 items reflecting disorganization and commotion. Parents will rate each item as true or false, with scores indicating higher or lower levels of chaos and disorganization.
Change in parenting | Change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured through the Coping with Children's Negative Emotions Scale (CCNES), a 12-item self-report measure of parental emotion parenting practices in response to children's expression of negative emotion. Responses are divided into six subscales representing six distinct types of parental responses. The responses will be grouped in two overall scores: Supportive (Expressive Encouragement, Problem-Focused, and Emotion-Focused Reactions) and Unsupportive (Punitive, Minimizing, and Distress Reactions) practices. Parents will rate the likelihood that they would respond in these distinct ways on a seven-point Likert scale from 1 (Very unlikely) to 7 (Very likely), with greater overall scores (range = 1-7) indicating greater levels of each type of parental response.
Change in child trauma symptoms | Change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured with the Child and Adolescent Trauma Screener (CATS), a 15-item screener of the occurrence of traumatic events, and 25-items of trauma symptoms. Parents will rate items on a four-point Likert scale from 0 (Never) to 3 (Almost always) with greater scores (range = 0 - 75) indicating more severe trauma symptoms.
Change in child positive and negative affect | Change at post-test (after completion of the waitlist or intervention treatment; an average range 4 - 6 months)
  This outcome will be measured with the Positive and Negative Affect Scale (PANAS), a 20-item questionnaire consisting of single-word items describing positive (e.g. excited) and negative (e.g. scared) feelings. Each item is rated on a 5-point scale (1 = Very slightly or not at all; 5 = Extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Kristel Thomassin, PhD, Principal Investigator — University of Guelph
Locations (2):
- Canada (2):
  - Maplewoods Centre for Family Therapy and Child Psychology, Guelph, Ontario
  - The Centre for Addition and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weisz JR, Kuppens S, Ng MY, Eckshtain D, Ugueto AM, Vaughn-Coaxum R, Jensen-Doss A, Hawley KM, Krumholz Marchette LS, Chu BC, Weersing VR, Fordwood SR. What five decades of research tells us about the effects of youth psychological therapy: A multilevel meta-analysis and implications for science and practice. Am Psychol. 2017 Feb-Mar;72(2):79-117. doi: 10.1037/a0040360. PMID 28221063
- [Background] Kreibig SD. Autonomic nervous system activity in emotion: a review. Biol Psychol. 2010 Jul;84(3):394-421. doi: 10.1016/j.biopsycho.2010.03.010. Epub 2010 Apr 4. PMID 20371374
- [Background] Sloan E, Hall K, Moulding R, Bryce S, Mildred H, Staiger PK. Emotion regulation as a transdiagnostic treatment construct across anxiety, depression, substance, eating and borderline personality disorders: A systematic review. Clin Psychol Rev. 2017 Nov;57:141-163. doi: 10.1016/j.cpr.2017.09.002. Epub 2017 Sep 11. PMID 28941927
- [Background] Fergusson DM, Woodward LJ. Mental health, educational, and social role outcomes of adolescents with depression. Arch Gen Psychiatry. 2002 Mar;59(3):225-31. doi: 10.1001/archpsyc.59.3.225. PMID 11879160
- [Background] Masten AS, Roisman GI, Long JD, Burt KB, Obradovic J, Riley JR, Boelcke-Stennes K, Tellegen A. Developmental cascades: linking academic achievement and externalizing and internalizing symptoms over 20 years. Dev Psychol. 2005 Sep;41(5):733-746. doi: 10.1037/0012-1649.41.5.733. PMID 16173871
- [Background] Masi G, Muratori P, Manfredi A, Lenzi F, Polidori L, Ruglioni L, Muratori F, Milone A. Response to treatments in youth with disruptive behavior disorders. Compr Psychiatry. 2013 Oct;54(7):1009-15. doi: 10.1016/j.comppsych.2013.04.007. Epub 2013 May 14. PMID 23683839
- [Background] Hollenstein T, McNeely A, Eastabrook J, Mackey A, Flynn J. Sympathetic and parasympathetic responses to social stress across adolescence. Dev Psychobiol. 2012 Mar;54(2):207-14. doi: 10.1002/dev.20582. Epub 2011 Jun 17. PMID 21688260
- [Background] Davis M, Thomassin K, Bilms J, Suveg C, Shaffer A, Beach SRH. Preschoolers' genetic, physiological, and behavioral sensitivity factors moderate links between parenting stress and child internalizing, externalizing, and sleep problems. Dev Psychobiol. 2017 May;59(4):473-485. doi: 10.1002/dev.21510. Epub 2017 Mar 14. PMID 28295263
- [Background] El-Sheikh M, Erath SA. Family conflict, autonomic nervous system functioning, and child adaptation: state of the science and future directions. Dev Psychopathol. 2011 May;23(2):703-21. doi: 10.1017/S0954579411000034. PMID 23786705
- [Background] McLaughlin KA, Alves S, Sheridan MA. Vagal regulation and internalizing psychopathology among adolescents exposed to childhood adversity. Dev Psychobiol. 2014 Jul;56(5):1036-51. doi: 10.1002/dev.21187. Epub 2013 Dec 11. PMID 24338154
- [Background] Lahey BB, Krueger RF, Rathouz PJ, Waldman ID, Zald DH. A hierarchical causal taxonomy of psychopathology across the life span. Psychol Bull. 2017 Feb;143(2):142-186. doi: 10.1037/bul0000069. Epub 2016 Dec 22. PMID 28004947
- [Background] Haltigan JD, Aitken M, Skilling T, Henderson J, Hawke L, Battaglia M, Strauss J, Szatmari P, Andrade BF. "P" and "DP:" Examining Symptom-Level Bifactor Models of Psychopathology and Dysregulation in Clinically Referred Children and Adolescents. J Am Acad Child Adolesc Psychiatry. 2018 Jun;57(6):384-396. doi: 10.1016/j.jaac.2018.03.010. Epub 2018 Apr 10. PMID 29859554
- [Background] Aitken M, Battaglia M, Marino C, Mahendran N, Andrade BF. Clinical utility of the CBCL Dysregulation Profile in children with disruptive behavior. J Affect Disord. 2019 Jun 15;253:87-95. doi: 10.1016/j.jad.2019.04.034. Epub 2019 Apr 9. PMID 31029857
- [Background] Bird HR, Canino GJ, Davies M, Ramirez R, Chavez L, Duarte C, Shen S. The Brief Impairment Scale (BIS): a multidimensional scale of functional impairment for children and adolescents. J Am Acad Child Adolesc Psychiatry. 2005 Jul;44(7):699-707. doi: 10.1097/01.chi.0000163281.41383.94. PMID 15968239
- [Background] Weisz JR, Vaughn-Coaxum RA, Evans SC, Thomassin K, Hersh J, Ng MY, Lau N, Lee EH, Raftery-Helmer JN, Mair P. Efficient Monitoring of Treatment Response during Youth Psychotherapy: The Behavior and Feelings Survey. J Clin Child Adolesc Psychol. 2020 Nov-Dec;49(6):737-751. doi: 10.1080/15374416.2018.1547973. Epub 2019 Jan 18. PMID 30657721
- [Background] Sachser C, Berliner L, Holt T, Jensen TK, Jungbluth N, Risch E, Rosner R, Goldbeck L. International development and psychometric properties of the Child and Adolescent Trauma Screen (CATS). J Affect Disord. 2017 Mar 1;210:189-195. doi: 10.1016/j.jad.2016.12.040. Epub 2016 Dec 27. PMID 28049104
- [Background] Lahey BB, Applegate B, Chronis AM, Jones HA, Williams SH, Loney J, Waldman ID. Psychometric characteristics of a measure of emotional dispositions developed to test a developmental propensity model of conduct disorder. J Clin Child Adolesc Psychol. 2008 Oct;37(4):794-807. doi: 10.1080/15374410802359635. PMID 18991130
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Buske-Kirschbaum A, Jobst S, Wustmans A, Kirschbaum C, Rauh W, Hellhammer D. Attenuated free cortisol response to psychosocial stress in children with atopic dermatitis. Psychosom Med. 1997 Jul-Aug;59(4):419-26. doi: 10.1097/00006842-199707000-00012. PMID 9251162
- [Background] Dickerson SS, Kemeny ME. Acute stressors and cortisol responses: a theoretical integration and synthesis of laboratory research. Psychol Bull. 2004 May;130(3):355-91. doi: 10.1037/0033-2909.130.3.355. PMID 15122924
- [Background] Helfinstein SM, Kirwan ML, Benson BE, Hardin MG, Pine DS, Ernst M, Fox NA. Validation of a child-friendly version of the monetary incentive delay task. Soc Cogn Affect Neurosci. 2013 Aug;8(6):720-6. doi: 10.1093/scan/nss057. Epub 2012 May 7. PMID 22569186
- [Background] Forbes EE, Hariri AR, Martin SL, Silk JS, Moyles DL, Fisher PM, Brown SM, Ryan ND, Birmaher B, Axelson DA, Dahl RE. Altered striatal activation predicting real-world positive affect in adolescent major depressive disorder. Am J Psychiatry. 2009 Jan;166(1):64-73. doi: 10.1176/appi.ajp.2008.07081336. Epub 2008 Dec 1. PMID 19047324
- [Background] Steinberg L. A Social Neuroscience Perspective on Adolescent Risk-Taking. Dev Rev. 2008 Mar;28(1):78-106. doi: 10.1016/j.dr.2007.08.002. PMID 18509515
- [Background] Silvers JA, Weber J, Wager TD, Ochsner KN. Bad and worse: neural systems underlying reappraisal of high- and low-intensity negative emotions. Soc Cogn Affect Neurosci. 2015 Feb;10(2):172-9. doi: 10.1093/scan/nsu043. Epub 2014 Mar 5. PMID 24603024
- [Background] Eisenberg N, Hofer C, Spinrad TL, Gershoff ET, Valiente C, Losoya SH, Zhou Q, Cumberland A, Liew J, Reiser M, Maxon E. Understanding mother-adolescent conflict discussions: concurrent and across-time prediction from youths' dispositions and parenting. Monogr Soc Res Child Dev. 2008;73(2):vii-viii, 1-160. doi: 10.1111/j.1540-5834.2008.00470.x. PMID 18702792
- [Background] Andreu Y, Galdon MJ, Dura E, Ferrando M, Murgui S, Garcia A, Ibanez E. Psychometric properties of the Brief Symptoms Inventory-18 (Bsi-18) in a Spanish sample of outpatients with psychiatric disorders. Psicothema. 2008 Nov;20(4):844-50. PMID 18940093
- [Background] Hallion LS, Steinman SA, Tolin DF, Diefenbach GJ. Psychometric Properties of the Difficulties in Emotion Regulation Scale (DERS) and Its Short Forms in Adults With Emotional Disorders. Front Psychol. 2018 Apr 19;9:539. doi: 10.3389/fpsyg.2018.00539. eCollection 2018. PMID 29725312
- [Background] Dumas JE, Nissley J, Nordstrom A, Smith EP, Prinz RJ, Levine DW. Home chaos: sociodemographic, parenting, interactional, and child correlates. J Clin Child Adolesc Psychol. 2005 Mar;34(1):93-104. doi: 10.1207/s15374424jccp3401_9. PMID 15677284
- [Background] Chorpita BF, Daleiden EL, Park AL, Ward AM, Levy MC, Cromley T, Chiu AW, Letamendi AM, Tsai KH, Krull JL. Child STEPs in California: A cluster randomized effectiveness trial comparing modular treatment with community implemented treatment for youth with anxiety, depression, conduct problems, or traumatic stress. J Consult Clin Psychol. 2017 Jan;85(1):13-25. doi: 10.1037/ccp0000133. Epub 2016 Aug 22. PMID 27548030
- [Background] Weisz JR, Chorpita BF, Palinkas LA, Schoenwald SK, Miranda J, Bearman SK, Daleiden EL, Ugueto AM, Ho A, Martin J, Gray J, Alleyne A, Langer DA, Southam-Gerow MA, Gibbons RD; Research Network on Youth Mental Health. Testing standard and modular designs for psychotherapy treating depression, anxiety, and conduct problems in youth: a randomized effectiveness trial. Arch Gen Psychiatry. 2012 Mar;69(3):274-82. doi: 10.1001/archgenpsychiatry.2011.147. Epub 2011 Nov 7. PMID 22065252
- [Background] McLeod BD, Weisz JR. The therapy process observational coding system-alliance scale: measure characteristics and prediction of outcome in usual clinical practice. J Consult Clin Psychol. 2005 Apr;73(2):323-33. doi: 10.1037/0022-006X.73.2.323. PMID 15796640
- [Background] Addis ME, Krasnow AD. A national survey of practicing psychologists' attitudes toward psychotherapy treatment manuals. J Consult Clin Psychol. 2000 Apr;68(2):331-9. doi: 10.1037//0022-006x.68.2.331. PMID 10780134

DOCUMENTS (2):
  • Study Protocol (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT05637320/Prot_003.pdf
  • Informed Consent Form (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/20/NCT05637320/ICF_002.pdf